CLINICAL TRIAL: NCT05404087
Title: Clinical Evaluation of Contrast Enhanced Breast CT to Improve Staging and Treatment Follow up in Women With Breast Cancer
Brief Title: Evaluation of Contrast Enhanced Breast CT for Diagnosis and Staging of Breast Cancer
Acronym: CEBCTvsMRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NL75855.091.21
Record Dates: First submitted 2022-05-24; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Pre-operative staging of breast cancer with CEBCT: Women who have been diagnosed with breast cancer and need to have a pre-operative staging and this will be done with contrast-enhanced breast CT.
  Interventions: Device: Dedicated breast CT
- Follow-up of women with breast cancer treated with neo-adjuvant chemotherapy: Women who are selected for neo-adjuvant chemotherapy to reduce the size of the tumor need to be followed-up in order to evaluate the treatment response.
  Interventions: Device: Dedicated breast CT

INTERVENTIONS:
Device: Dedicated breast CT — Administration of contrast agent and scanning of the breast in order to evaluate the enhancement of the tumor

SUMMARY:
Contrast-enhanced breast CT is a novel high resolution and fully 3D imaging method to document abnormalities within the breast. I will establish its value for breast cancer staging and in monitoring therapy response.

DETAILED DESCRIPTION:
Breast CT is a novel modality that has not been largely evaluated in a clinical setting. Only recently FDA and CE marked BCT machines have been released, and the number of installed bases internationally is below 10 (although rapidly rising).

Internationally only a few studies on contrast enhanced breast CT have been performed in small numbers of patients, albeit with excellent results. Nevertheless, substantial evidence for this novel modality is still absent. In particular, the correlation of enhancement and histological grade of DCIS, correlation of CEBCT findings with histopathology, and prediction and assessment of primary systemic treatment are open fields for which more substantial evaluation is clearly needed. In this study we want to establish the value of CEBCT in staging of women with breast cancer, particularly those with extensive carcinoma in situ (DCIS), and in the evaluation of women treated with primary systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of breast cancer
* Scheduled for a pre-surgery staging contrast enhanced breast MRI
* Eligible for primary systemic therapy

Exclusion Criteria:

* Women with suspected or confirmed pregnancy
* Women with prior history of breast cancer
* Women who are breastfeeding
* Women who are very frail and unable to cooperate
* Women who cannot give informed consent
* Contra indication of iodine contrast (i.e. untreatable contrast allergy, renal function impairment (GFR <60 ml/min/1.73m2))
* Contra indication for irradiation (i.e. genetic mutation that predispose to breast cancer)
* Male subjects

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer
Sampling Method: Probability Sample
Enrollment: 413 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of CEBCT error rate vs DCE MRI error rate, both as compared to the golden standard for tumor staging. | 3 years
  Non-inferiority of CEBCT error rate against the golden standard, i.e. histopathology, to DCE MRI error rate against the golden standard for tumor staging.
  i.e. histopathology, to DCE MRI error rate against the golden standard for tumor staging.
Non-inferiority of CEBCT to predict pCR after primary systemic therapy as compared to DCE MRI. | 3 years
  Non-inferiority of CEBCT to predict pCR after primary systemic therapy as compared to DCE MRI computed from the area under the receiver operating characteristic (ROC) curve (AUC) (or AUROC).

SECONDARY OUTCOMES:
Concordance of tumor extent between CEBCT and large section histopathology | 3 years
  We will evaluate the rate of concordance between the size of the tumour determined at CEBCT images and those at final histopathology sections
Frequency of detection of contralateral cancers with CEBCT | 3 years
  We will record how many times we will find a contralateral incidental breast cancer, not previously reported, after performing CEBCT
Concordance between morphological and enhancement characteristics of cancers on CEBCT to their expected response to primary systemic therapy. | 3 years
  We will evaluate the rate of concordance of breast cancer response to primary systemic therapy compared to the expected response based on literature by evaluating their morphological and enhancement characteristics at CEBCT examinations
Potential of CEBCT predicting the response to primary systemic therapy early in treatment | 3 years
  We will assess the potential of CEBCT in predicting the response of breast cancer to primary systemic therapy as compared to the assessment made at final histopathology section

CONTACTS AND LOCATIONS:
Overall Officials: Ritse Mann, MD-PhD, Principal Investigator — Radboudumc/The Netherlands Cancer Institute

IPD SHARING:
Plan to Share IPD: Undecided
We will evaluate the possibility to share anonimised data for future research

DOCUMENTS (1):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT05404087/Prot_000.pdf